CLINICAL TRIAL: NCT02979535
Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Cervarix® in Healthy Female Subjects Aged 9 to 14 Years in Mexico
Brief Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Cervarix®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYD71; U1111-1161-3455 (Other: WHO); 2019-000994-22 (EudraCT Number)
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Human Papillomavirus Disease
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; Human Papillomavirus Disease; CYD Dengue Vaccine; Dengvaxia®; Cervarix®
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Dengue Vaccines; human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CYD Dengue Vaccine + Cervarix (Concomitant Administration) (Experimental): Participants received 3 doses of CYD dengue vaccine 0.5 milliliter (mL) subcutaneously (SC) at Day 0, Month 6, and Month 12 and 2 doses of Cervarix vaccine 0.5 mL Intramuscularly (IM) concomitantly with the 2 first doses of CYD dengue vaccine.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Human Papillomavirus Bivalent [Types 16 and 18] Vaccine, Recombinant
- CYD Dengue Vaccine + Cervarix (Sequential Administration) (Experimental): Participants received 3 doses of CYD dengue vaccine 0.5 mL SC at Month 1, Month 7, and Month 13 along with the 2 doses of Cervarix vaccine 0.5 mL IM at Day 0 and Month 6 sequentially (i.e., one month before) to each of the 2 first doses of CYD dengue vaccine.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Human Papillomavirus Bivalent [Types 16 and 18] Vaccine, Recombinant

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 mL, SC at Day 0, Months 6 and 12
  Other Names: Dengvaxia®
  Arms: CYD Dengue Vaccine + Cervarix (Concomitant Administration)
Biological: CYD Dengue Vaccine — 0.5 mL, SC at Months 1, 7, and 13
  Other Names: Dengvaxia®
  Arms: CYD Dengue Vaccine + Cervarix (Sequential Administration)
Biological: Human Papillomavirus Bivalent [Types 16 and 18] Vaccine, Recombinant — 0.5 mL, IM at Day 0 and Month 6
  Other Names: Cervarix®
  Arms: CYD Dengue Vaccine + Cervarix (Concomitant Administration)
Biological: Human Papillomavirus Bivalent [Types 16 and 18] Vaccine, Recombinant — 0.5 mL, IM at Day 0 and Month 6
  Other Names: Cervarix®
  Arms: CYD Dengue Vaccine + Cervarix (Sequential Administration)

SUMMARY:
The aim of this study was to investigate the immunogenicity and safety of CYD dengue vaccine and Cervarix when administered concomitantly or sequentially in healthy female participants aged 9-14 years of age.

Primary objectives:

* To demonstrate that the humoral immune response (in terms of geometric mean titers [GMTs]) to Cervarix after concomitant administration with the CYD dengue vaccine is non-inferior to the humoral immune response (in terms of GMTs) after sequential administration with the CYD dengue vaccine measured 28 days after the last dose of Cervarix.
* To demonstrate that the humoral immune response (in terms of GMTs) to the CYD dengue vaccine after concomitant administration with Cervarix is non-inferior to the humoral immune response (in terms of GMTs) to the CYD dengue vaccine after sequential administration with Cervarix measured 28 days after the last dose of the CYD dengue vaccine.

Secondary Objectives:

* To demonstrate that the humoral immune response (in terms of seroconversion) to Cervarix after concomitant administration with the CYD dengue vaccine is non-inferior to the humoral immune response (in terms of seroconversion) to Cervarix sequential administration with the CYD dengue vaccine measured 28 days after the last dose of Cervarix.
* To describe the humoral immune response to Cervarix at baseline and after each dose of Cervarix in each and any group.
* To describe the humoral immune response to the CYD dengue vaccine at baseline and after each dose of the CYD dengue vaccine, in each and any group.
* To describe the safety of Cervarix and CYD dengue vaccine after each and any dose in each group.

DETAILED DESCRIPTION:
Participants received 3 doses of the CYD dengue vaccine and 2 doses of Cervarix administered either concomitantly or sequentially. Due to a protocol amendment, only previously dengue exposed participants (seropositive for dengue before vaccination) were eligible to complete the vaccination schedule and be assessed for CYD immunogenicity and human papilloma virus (HPV) immunogenicity. Dengue unexposed participants (seronegative for dengue before vaccination) did not receive the third CYD dengue vaccine injection, but were followed for safety up to 6 months after the last injection.

Safety assessments included solicited reactions within 7 or 14 days after each injection, unsolicited adverse events within 28 days after each injection, and serious adverse events during the study period. All participants were included in the assessment of safety up to 6 months after the last injection.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 9 to 14 years (i.e., from the day of the 9th birthday to the day prior to the 15th birthday) on the day of inclusion.
* Informed consent form (ICF) or Assent form (AF) had been signed and dated by the participant (based on local regulations), and/or ICF had been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* Participant (or participant and parent[s] or another legally acceptable representative) was (were) able to attend all scheduled visits and complied with all trial procedures.
* Participant in good health, based on medical history, and physical examination.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Previous vaccination against dengue disease with the trial vaccine.
* Previous vaccination against HPV disease with either the trial vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency (including HIV infection with impaired immune function); or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of HPV infection, confirmed either clinically, serologically, or microbiologically as reported by participant or parent(s) or another legally acceptable representative.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia, contraindicating IM vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that, based on investigator's judgment, might interfere with the participant's ability to comply with trial procedures.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Identified as an Investigator or employee of the Investigator with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Self-reported Hepatitis B, Hepatitis C infection.

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Arredondo JL, Villagomez Martinez SM, Concepcion Morales M, Meyer S, Toh ML, Zocchetti C, Vigne C, Mascarenas C. Immunogenicity and safety of a tetravalent dengue vaccine and a bivalent HPV vaccine given concomitantly or sequentially in girls aged 9 to 14 years in Mexico. Vaccine. 2021 Jun 8;39(25):3388-3396. doi: 10.1016/j.vaccine.2021.04.064. Epub 2021 May 13. PMID 33992441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 16 November 2016 to 13 March 2017 at 3 centers in Mexico.
Pre-assignment Details: A total of 480 participants were enrolled and randomized in this study.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Started | 239 | 241
Safety Analysis Set (Safety analysis set was defined as participants who had received at least 1 dose of study vaccines.) | 237 | 241
Completed | 144 | 140
Not Completed | 95 | 101
Not completed — Non compliance with the protocol | 78 | 82
Not completed — Consent withdrawn by participant | 11 | 18
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed on all randomized population which included participants for whom an injection group were allocated.
Groups:
- CYD Dengue Vaccine + Cervarix (Concomitant Administration): Participants received 3 doses of CYD dengue vaccine 0.5 mL SC at Day 0, Month 6, and Month 12 and 2 doses of Cervarix vaccine 0.5 mL IM concomitantly with the 2 first doses of CYD dengue vaccine.
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration) | Total
Number analyzed (Participants) | 239 | 241 | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.50 (1.00) | 9.56 (1.05) | 9.53 (1.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 241 | 480
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Not reported | 239 | 241 | 480

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) Against Each Cervarix Human Papillomavirus (HPV) Antigen (HPV-16 and HPV-18) 28 Days After Last Cervarix Vaccination in the Previously Dengue Seropositive Participants
Description: GMTs against each Cervarix HPV antigen (HPV-16 and HPV-18) were assessed using an enzyme-linked immunosorbent assay (ELISA) method. Dengue seropositive participants at baseline were defined as those participants with titers greater than or equal to (>=) 10 (1/dilutions [dil]) for at least one serotype with the parental dengue virus strain.
Time Frame: 28 days after the last Cervarix vaccination
Population: Analysis was performed on per-protocol analysis set (PPS) for Cervarix which included participants who received at least one dose of Cervarix vaccine and had no relevant protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Endotoxin Units per milliliter (EU/mL)
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 118 | 114
Endotoxin Units per milliliter (EU/mL)
  HPV-16 | 2149 [1877 to 2460] | 2268 [1946 to 2644]
  HPV-18 | 833 [727 to 954] | 845 [723 to 987]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine + Cervarix (Concomitant Administration) vs CYD Dengue Vaccine + Cervarix (Sequential Administration); Antigen HPV-16; Test type: Other; GMT ratio = 0.947, 95% CI 2-sided [0.773 to 1.16]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine + Cervarix (Concomitant Administration) vs CYD Dengue Vaccine + Cervarix (Sequential Administration); Antigen HPV-18; Test type: Other; GMT ratio = 0.986, 95% CI 2-sided [0.803 to 1.21]

2. Primary Outcome: GMTs Against Each Dengue Virus Serotype 28 Days After the Third CYD Dengue Vaccination in the Previously Dengue Seropositive Participants
Description: The GMTs against each of the four parental dengue virus serotypes (Serotypes 1, 2, 3, and 4) of CYD dengue vaccine were assessed using the 50% plaque reduction neutralization test (PRNT50) assay. Dengue seropositive participants at baseline were defined as those participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strain.
Time Frame: 28 days after third CYD dengue vaccination
Population: Analysis was performed on the full analysis set (FAS) which was defined as the subset of participants who received at least one dose of the study vaccine. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer (1/dilution)
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 143 | 140
titer (1/dilution)
  Serotype 1 | 384 [291 to 507] | 393 [292 to 528]
  Serotype 2 | 670 [535 to 839] | 735 [575 to 940]
  Serotype 3 | 357 [305 to 418] | 388 [325 to 463]
  Serotype 4 | 247 [213 to 287] | 265 [220 to 320]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine + Cervarix (Concomitant Administration) vs CYD Dengue Vaccine + Cervarix (Sequential Administration); Dengue Virus Serotype 1; Test type: Other; GMT ratio = 0.977, 95% CI 2-sided [0.653 to 1.46]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine + Cervarix (Concomitant Administration) vs CYD Dengue Vaccine + Cervarix (Sequential Administration); Dengue Virus Serotype 2; Test type: Other; GMT ratio = 0.911, 95% CI 2-sided [0.654 to 1.27]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine + Cervarix (Concomitant Administration) vs CYD Dengue Vaccine + Cervarix (Sequential Administration); Dengue Virus Serotype 3; Test type: Other; GMT ratio = 0.921, 95% CI 2-sided [0.727 to 1.17]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine + Cervarix (Concomitant Administration) vs CYD Dengue Vaccine + Cervarix (Sequential Administration); Dengue Virus Serotype 4; Test type: Other; GMT ratio = 0.931, 95% CI 2-sided [0.733 to 1.18]

3. Secondary Outcome: GMTs Against Each Cervarix HPV Antigen (HPV-16 and HPV-18) at Day 0 and 28 Days After Each Cervarix Vaccination in the Previously Dengue Seropositive Participants
Description: The GMTs against each Cervarix HPV antigen (HPV-16 and HPV-18) were assessed using an ELISA method. Dengue seropositive participants at baseline were defined as those participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strain.
Time Frame: Day 0 and 28 days after each Cervarix vaccination
Population: Analysis was performed on FAS population. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants with available data for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 154 | 151
EU/mL
  HPV-16: Day 0 | 1.61 [1.31 to 1.97] | 1.58 [1.29 to 1.93]
  HPV-16: 28 days post vaccination 1: number analyzed (Participants) | 150 | 151
  HPV-16: 28 days post vaccination 1 | 118 [98.7 to 142] | 140 [116 to 170]
  HPV-16: 28 days post vaccination 2: number analyzed (Participants) | 149 | 147
  HPV-16: 28 days post vaccination 2 | 2089 [1852 to 2356] | 2162 [1869 to 2501]
  HPV-18: Day 0 | 1.34 [1.15 to 1.55] | 1.34 [1.16 to 1.54]
  HPV-18: 28 days post vaccination 1: number analyzed (Participants) | 150 | 151
  HPV-18: 28 days post vaccination 1 | 53.8 [44.1 to 65.7] | 68.6 [56.5 to 83.4]
  HPV-18: 28 days post vaccination 2: number analyzed (Participants) | 149 | 147
  HPV-18: 28 days post vaccination 2 | 846 [752 to 951] | 846 [728 to 984]

4. Secondary Outcome: Percentage of Participants With Seroconversion Against Each Cervarix HPV Antigen (HPV-16 and HPV-18) 28 Days After Each Dose of Cervarix Vaccination in the Previously Dengue Seropositive Participants
Description: Neutralizing antibodies against each Cervarix HPV antigen (HPV-16 and HPV-18) were assessed using an ELISA method. Seroconversion was defined as changing serostatus from seronegative at baseline to seropositive (greater than [>] lower limit of quantitation [LLOQ] of the assay) or >=4-fold rise in antibody titer if seropositive at baseline (i.e., at least one antibody levels against Cervarix HPV antigens > LLOQ at baseline). The LLOQ for HPV-16 and HPV-18 was less than (<) 2.0 International Units per milliliter (IU/mL).
Time Frame: 28 days after each Cervarix vaccination
Population: Analysis was performed on FAS population. Here, "overall number of participants" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants with available data for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 154 | 151
percentage of participants
  HPV-16: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 151
  HPV-16: 28 days post-vaccination 1 | 98.0 [94.3 to 99.6] | 99.3 [96.4 to 100.0]
  HPV-16: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 147
  HPV-16: 28 days post-vaccination 2 | 98.7 [95.2 to 99.8] | 99.3 [96.3 to 100.0]
  HPV-18: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 151
  HPV-18: 28 days post-vaccination 1 | 100.0 [97.6 to 100.0] | 98.7 [95.3 to 99.8]
  HPV-18: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 147
  HPV-18: 28 days post-vaccination 2 | 99.3 [96.3 to 100.0] | 100.0 [97.5 to 100.0]

5. Secondary Outcome: GMTs Against Each Dengue Virus Serotype of CYD Dengue Vaccine at Day 0 and 28 Days After Each Dose of CYD Dengue Vaccination in the Previously Dengue Seropositive Participants
Description: The GMTs against each of the four parental dengue virus serotypes (Serotypes 1, 2, 3, and 4) of CYD dengue vaccine were assessed using the PRNT50 assay. Dengue seropositive participants at baseline were defined as those participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strain.
Time Frame: Day 0 and 28 days after each CYD dengue vaccine vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer (1/dilution)
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 154 | 151
titer (1/dilution)
  Serotype 1: Day 0 | 150 [99.7 to 225] | 108 [72.1 to 163]
  Serotype 1: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 1: 28 days post-vaccination 1 | 711 [498 to 1016] | 586 [409 to 840]
  Serotype 1: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 1: 28 days post-vaccination 2 | 460 [336 to 630] | 476 [337 to 674]
  Serotype 1: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 1: 28 days post-vaccination 3 | 384 [291 to 507] | 393 [292 to 528]
  Serotype 2: Day 0 | 193 [141 to 263] | 188 [135 to 262]
  Serotype 2: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 2: 28 days post-vaccination 1 | 1168 [879 to 1552] | 1163 [847 to 1597]
  Serotype 2: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 2: 28 days post-vaccination 2 | 618 [492 to 776] | 703 [541 to 913]
  Serotype 2: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 2: 28 days post-vaccination 3 | 670 [535 to 839] | 735 [575 to 940]
  Serotype 3: Day 0 | 98.5 [72.2 to 135] | 90.2 [67.2 to 121]
  Serotype 3: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 3: 28 days post-vaccination 1 | 499 [386 to 644] | 503 [385 to 656]
  Serotype 3: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 3: 28 days post-vaccination 2 | 299 [251 to 358] | 361 [294 to 445]
  Serotype 3: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 3: 28 days post-vaccination 3 | 357 [305 to 418] | 388 [325 to 463]
  Serotype 4: Day 0 | 47.1 [34.6 to 64.0] | 38.0 [28.4 to 50.9]
  Serotype 4: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 4: 28 days post-vaccination 1 | 423 [336 to 532] | 449 [365 to 552]
  Serotype 4: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 4: 28 days post-vaccination 2 | 267 [225 to 316] | 262 [219 to 314]
  Serotype 4: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 4: 28 days post-vaccination 3 | 247 [213 to 287] | 265 [220 to 320]

6. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers >=10 (1/Dil) Against Each of the 4 Dengue Virus Serotypes of CYD Dengue Vaccine at Day 0 And 28 Days After Each Dose of CYD Dengue Vaccination in the Previously Dengue Seropositive Participants
Description: Dengue neutralizing antibody levels against each of the 4 dengue virus serotypes (Serotypes 1, 2, 3, and 4) were measured by PRNT50. Dengue seropositive participants at baseline were defined as those participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strain.
Time Frame: Day 0 and 28 days after each CYD dengue vaccine vaccination
Population: Analysis was performed on FAS population. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants with available data for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 154 | 151
percentage of participants
  Serotype 1: Day 0 | 74.0 [66.4 to 80.8] | 68.9 [60.8 to 76.2]
  Serotype 1: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 1: 28 days post-vaccination 1 | 94.7 [89.8 to 97.7] | 95.3 [90.5 to 98.1]
  Serotype 1: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 1: 28 days post-vaccination 2 | 97.3 [93.3 to 99.3] | 97.3 [93.1 to 99.2]
  Serotype 1: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 1: 28 days post-vaccination 3 | 99.3 [96.2 to 100.0] | 97.9 [93.9 to 99.6]
  Serotype 2: Day 0 | 92.9 [87.6 to 96.4] | 91.4 [85.7 to 95.3]
  Serotype 2: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 2: 28 days post-vaccination 1 | 96.7 [92.4 to 98.9] | 93.9 [88.8 to 97.2]
  Serotype 2: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 2: 28 days post-vaccination 2 | 100.0 [97.6 to 100.0] | 98.6 [95.1 to 99.8]
  Serotype 2: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 2: 28 days post-vaccination 3 | 100.0 [97.5 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 3: Day 0 | 82.5 [75.5 to 88.1] | 83.4 [76.5 to 89.0]
  Serotype 3: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 3: 28 days post-vaccination 1 | 96.7 [92.4 to 98.9] | 96.6 [92.3 to 98.9]
  Serotype 3: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 3: 28 days post-vaccination 2 | 99.3 [96.3 to 100.0] | 100.0 [97.5 to 100.0]
  Serotype 3: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 3: 28 days post-vaccination 3 | 99.3 [96.2 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 4: Day 0 | 68.8 [60.9 to 76.0] | 66.9 [58.8 to 74.3]
  Serotype 4: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  Serotype 4: 28 days post-vaccination 1 | 97.3 [93.3 to 99.3] | 98.6 [95.2 to 99.8]
  Serotype 4: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  Serotype 4: 28 days post-vaccination 2 | 100.0 [97.6 to 100.0] | 100.0 [97.5 to 100.0]
  Serotype 4: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  Serotype 4: 28 days post-vaccination 3 | 100.0 [97.5 to 100.0] | 98.6 [94.9 to 99.8]

7. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers >=10 (1/Dil) Against At Least 1,2,3,or4 Dengue Virus Serotypes of CYD Dengue Vaccine at Day 0 And 28 Days After Each Dose of CYD Dengue Vaccination in Previously Dengue Seropositive Participants
Description: as for outcome 6
Time Frame: Day 0 and 28 days after each CYD dengue vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 154 | 151
percentage of participants
  At least 1 Serotype: Day 0 | 100.0 [97.6 to 100.0] | 100.0 [97.6 to 100.0]
  At least 1 Serotype: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  At least 1 Serotype: 28 days post-vaccination 1 | 99.3 [96.3 to 100.0] | 99.3 [96.3 to 100.0]
  At least 1 Serotype: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  At least 1 Serotype: 28 days post-vaccination 2 | 100.0 [97.6 to 100.0] | 100.0 [97.5 to 100.0]
  At least 1 Serotype: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  At least 1 Serotype: 28 days post-vaccination 3 | 100.0 [97.5 to 100.0] | 100.0 [97.4 to 100.0]
  At least 2 Serotype: Day 0 | 84.4 [77.7 to 89.8] | 82.8 [75.8 to 88.4]
  At least 2 Serotype: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  At least 2 Serotype: 28 days post-vaccination 1 | 98.0 [94.3 to 99.6] | 98.0 [94.2 to 99.6]
  At least 2 Serotype: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  At least 2 Serotype: 28 days post-vaccination 2 | 100.0 [97.6 to 100.0] | 100.0 [97.5 to 100.0]
  At least 2 Serotype: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  At least 2 Serotype: 28 days post-vaccination 3 | 100.0 [97.5 to 100.0] | 100.0 [97.4 to 100.0]
  At least 3 Serotype: Day 0 | 74.0 [66.4 to 80.8] | 72.8 [65.0 to 79.8]
  At least 3 Serotype: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  At least 3 Serotype: 28 days post-vaccination 1 | 95.3 [90.6 to 98.1] | 94.6 [89.6 to 97.6]
  At least 3 Serotype: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  At least 3 Serotype: 28 days post-vaccination 2 | 99.3 [96.3 to 100.0] | 98.6 [95.1 to 99.8]
  At least 3 Serotype: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  At least 3 Serotype: 28 days post-vaccination 3 | 100.0 [97.5 to 100.0] | 98.6 [94.9 to 99.8]
  All 4 Serotypes: Day 0 | 59.7 [51.5 to 67.6] | 55.0 [46.7 to 63.1]
  All 4 Serotypes: 28 days post-vaccination 1: number analyzed (Participants) | 150 | 148
  All 4 Serotypes: 28 days post-vaccination 1 | 92.7 [87.3 to 96.3] | 92.6 [87.1 to 96.2]
  All 4 Serotypes: 28 days post-vaccination 2: number analyzed (Participants) | 149 | 146
  All 4 Serotypes: 28 days post-vaccination 2 | 97.3 [93.3 to 99.3] | 97.3 [93.1 to 99.2]
  All 4 Serotypes: 28 days post-vaccination 3: number analyzed (Participants) | 143 | 140
  All 4 Serotypes: 28 days post-vaccination 3 | 98.6 [95.0 to 99.8] | 97.9 [93.9 to 99.6]

8. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers Above Pre-defined Thresholds Against Each Dengue Virus Serotypes of CYD at Baseline And 28 Days After Each Dose of CYD Dengue Vaccination in Dengue Seropositive Participants
Description: Dengue neutralizing antibody levels against each of the 4 dengue virus serotypes (Serotypes 1, 2, 3, and 4) were measured by PRNT50. Dengue seropositive participants at baseline were defined as those participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strain. Percentage of participants with neutralizing antibody titers above pre-defined thresholds (<10, >=10 and >=100 [1/dil]) against each dengue virus serotypes of CYD were reported.
Time Frame: Day 0 and 28 days after each CYD dengue vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 154 | 151
percentage of participants
  Serotype 1: Pre-vaccination 1 <10 (1/dil) | 26.0 [19.2 to 33.6] | 31.1 [23.8 to 39.2]
  Serotype 1: Pre-vaccination 1 >=10 (1/dil) | 74.0 [66.4 to 80.8] | 68.9 [60.8 to 76.2]
  Serotype 1: Pre-vaccination 1 >=100 (1/dil) | 61.0 [52.9 to 68.8] | 56.3 [48.0 to 64.3]
  Serotype 1: Post-vaccination 1 <10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 1: Post-vaccination 1 <10 (1/dil) | 5.3 [2.3 to 10.2] | 4.7 [1.9 to 9.5]
  Serotype 1: Post-vaccination 1 >=10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 1: Post-vaccination 1 >=10 (1/dil) | 94.7 [89.8 to 97.7] | 95.3 [90.5 to 98.1]
  Serotype 1: Post-vaccination 1 >=100 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 1: Post-vaccination 1 >=100 (1/dil) | 82.0 [74.9 to 87.8] | 78.4 [70.9 to 84.7]
  Serotype 1: Post-vaccination 2 <10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 1: Post-vaccination 2 <10 (1/dil) | 2.7 [0.7 to 6.7] | 2.7 [0.8 to 6.9]
  Serotype 1: Post-vaccination 2 >=10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 1: Post-vaccination 2 >=10 (1/dil) | 97.3 [93.3 to 99.3] | 97.3 [93.1 to 99.2]
  Serotype 1: Post-vaccination 2 >=100 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 1: Post-vaccination 2 >=100 (1/dil) | 77.2 [69.6 to 83.7] | 72.6 [64.6 to 79.7]
  Serotype 1: Post-vaccination 3 <10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 1: Post-vaccination 3 <10 (1/dil) | 0.7 [0.0 to 3.8] | 2.1 [0.4 to 6.1]
  Serotype 1: Post-vaccination 3 >=10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 1: Post-vaccination 3 >=10 (1/dil) | 99.3 [96.2 to 100.0] | 97.9 [93.9 to 99.6]
  Serotype 1: Post-vaccination 3 >=100 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 1: Post-vaccination 3 >=100 (1/dil) | 74.8 [66.9 to 81.7] | 76.4 [68.5 to 83.2]
  Serotype 2: Pre-vaccination 1 <10 (1/dil) | 7.1 [3.6 to 12.4] | 8.6 [4.7 to 14.3]
  Serotype 2: Pre-vaccination 1 >=10 (1/dil) | 92.9 [87.6 to 96.4] | 91.4 [85.7 to 95.3]
  Serotype 2: Pre-vaccination 1 >=100 (1/dil) | 59.1 [50.9 to 66.9] | 61.6 [53.3 to 69.4]
  Serotype 2: Post-vaccination 1 <10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 2: Post-vaccination 1 <10 (1/dil) | 3.3 [1.1 to 7.6] | 6.1 [2.8 to 11.2]
  Serotype 2: Post-vaccination 1 >=10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 2: Post-vaccination 1 >=10 (1/dil) | 96.7 [92.4 to 98.9] | 93.9 [88.8 to 97.2]
  Serotype 2: Post-vaccination 1 >=100 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 2: Post-vaccination 1 >=100 (1/dil) | 91.3 [85.6 to 95.3] | 91.9 [86.3 to 95.7]
  Serotype 2: Post-vaccination 2 <10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 2: Post-vaccination 2 <10 (1/dil) | 0.0 [0.0 to 2.4] | 1.4 [0.2 to 4.9]
  Serotype 2: Post-vaccination 2 >=10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 2: Post-vaccination 2 >=10 (1/dil) | 100.0 [97.6 to 100.0] | 98.6 [95.1 to 99.8]
  Serotype 2: Post-vaccination 2 >=100 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 2: Post-vaccination 2 >=100 (1/dil) | 90.6 [84.7 to 94.8] | 90.4 [84.4 to 94.7]
  Serotype 2: Post-vaccination 3 <10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 2: Post-vaccination 3 <10 (1/dil) | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.6]
  Serotype 2: Post-vaccination 3 >=10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 2: Post-vaccination 3 >=10 (1/dil) | 100.0 [97.5 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 2: Post-vaccination 3 >=100 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 2: Post-vaccination 3 >=100 (1/dil) | 95.1 [90.2 to 98.0] | 90.7 [84.6 to 95.0]
  Serotype 3: Pre-vaccination 1 <10 (1/dil) | 17.5 [11.9 to 24.5] | 16.6 [11.0 to 23.5]
  Serotype 3: Pre-vaccination 1 >=10 (1/dil) | 82.5 [75.5 to 88.1] | 83.4 [76.5 to 89.0]
  Serotype 3: Pre-vaccination 1 >=100 (1/dil) | 51.3 [43.1 to 59.4] | 49.0 [40.8 to 57.3]
  Serotype 3: Post-vaccination 1 <10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 3: Post-vaccination 1 <10 (1/dil) | 3.3 [1.1 to 7.6] | 3.4 [1.1 to 7.7]
  Serotype 3: Post-vaccination 1 >=10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 3: Post-vaccination 1 >=10 (1/dil) | 96.7 [92.4 to 98.9] | 96.6 [92.3 to 98.9]
  Serotype 3: Post-vaccination 1 >=100 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 3: Post-vaccination 1 >=100 (1/dil) | 88.7 [82.5 to 93.3] | 87.8 [81.5 to 92.6]
  Serotype 3: Post-vaccination 2 <10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 3: Post-vaccination 2 <10 (1/dil) | 0.7 [0.0 to 3.7] | 0.0 [0.0 to 2.5]
  Serotype 3: Post-vaccination 2 >=10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 3: Post-vaccination 2 >=10 (1/dil) | 99.3 [96.3 to 100.0] | 100.0 [97.5 to 100.0]
  Serotype 3: Post-vaccination 2 >=100 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 3: Post-vaccination 2 >=100 (1/dil) | 87.2 [80.8 to 92.1] | 87.0 [80.4 to 92.0]
  Serotype 3: Post-vaccination 3 <10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 3: Post-vaccination 3 <10 (1/dil) | 0.7 [0.0 to 3.8] | 0.0 [0.0 to 2.6]
  Serotype 3: Post-vaccination 3 >=10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 3: Post-vaccination 3 >=10 (1/dil) | 99.3 [96.2 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 3: Post-vaccination 3 >=100 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 3: Post-vaccination 3 >=100 (1/dil) | 94.4 [89.3 to 97.6] | 90.7 [84.6 to 95.0]
  Serotype 4: Pre-vaccination 1 <10 (1/dil) | 31.2 [24.0 to 39.1] | 33.1 [25.7 to 41.2]
  Serotype 4: Pre-vaccination 1 >=10 (1/dil) | 68.8 [60.9 to 76.0] | 66.9 [58.8 to 74.3]
  Serotype 4: Pre-vaccination 1 >=100 (1/dil) | 33.1 [25.8 to 41.1] | 29.8 [22.6 to 37.8]
  Serotype 4: Post-vaccination 1 <10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 4: Post-vaccination 1 <10 (1/dil) | 2.7 [0.7 to 6.7] | 1.4 [0.2 to 4.8]
  Serotype 4: Post-vaccination 1 >=10 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 4: Post-vaccination 1 >=10 (1/dil) | 97.3 [93.3 to 99.3] | 98.6 [95.2 to 99.8]
  Serotype 4: Post-vaccination 1 >=100 (1/dil): number analyzed (Participants) | 150 | 148
  Serotype 4: Post-vaccination 1 >=100 (1/dil) | 87.3 [80.9 to 92.2] | 89.9 [83.8 to 94.2]
  Serotype 4: Post-vaccination 2 <10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 4: Post-vaccination 2 <10 (1/dil) | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 2.5]
  Serotype 4: Post-vaccination 2 >=10 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 4: Post-vaccination 2 >=10 (1/dil) | 100.0 [97.6 to 100.0] | 100.0 [97.5 to 100.0]
  Serotype 4: Post-vaccination 2 >=100 (1/dil): number analyzed (Participants) | 149 | 146
  Serotype 4: Post-vaccination 2 >=100 (1/dil) | 82.6 [75.5 to 88.3] | 80.1 [72.7 to 86.3]
  Serotype 4: Post-vaccination 3 <10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 4: Post-vaccination 3 <10 (1/dil) | 0.0 [0.0 to 2.5] | 1.4 [0.2 to 5.1]
  Serotype 4: Post-vaccination 3 >=10 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 4: Post-vaccination 3 >=10 (1/dil) | 100.0 [97.5 to 100.0] | 98.6 [94.9 to 99.8]
  Serotype 4: Post-vaccination 3 >=100 (1/dil): number analyzed (Participants) | 143 | 140
  Serotype 4: Post-vaccination 3 >=100 (1/dil) | 83.2 [76.1 to 88.9] | 83.6 [76.4 to 89.3]

9. Secondary Outcome: Number of Participants Reporting Immediate Adverse Events (AEs) Following Vaccination With Cervarix or CYD Dengue Vaccine
Description: Any unsolicited systemic AE occurred during the first 30 minutes post-vaccination was recorded on the case report form (CRF) as immediate AE.
Time Frame: Within 30 minutes after each and any vaccination
Population: Analysis was performed on safety analysis set which included those participants who had received at least one dose of the study vaccines. Here, "number analyzed" signifies participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 237 | 241
Participants
  After any CYD/Cervarix vaccination | 0 | 0
  Post CYD/Cervarix vaccination 1 | 0 | 0
  Post CYD/Cervarix vaccination 2: number analyzed (Participants) | 227 | 229
  Post CYD/Cervarix vaccination 2 | 0 | 0
  Post CYD vaccination 3: number analyzed (Participants) | 145 | 141
  Post CYD vaccination 3 | 0 | 0

10. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions Following Vaccination With Cervarix or CYD Dengue Vaccine
Description: Solicited injection site reactions included pain, erythema, and swelling.
Time Frame: Up to 7 days after each and any vaccination
Population: Analysis was performed on safety analysis set. Here, "number analyzed" signifies participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 237 | 241
Participants
  Pain: Post any CYD/Cervarix vaccine: number analyzed (Participants) | 231 | 234
  Pain: Post any CYD/Cervarix vaccine | 212 | 221
  Pain: Post CYD/Cervarix vaccination 1: number analyzed (Participants) | 231 | 234
  Pain: Post CYD/Cervarix vaccination 1 | 202 | 206
  Pain: Post CYD/Cervarix vaccination 2: number analyzed (Participants) | 226 | 229
  Pain: Post CYD/Cervarix vaccination 2 | 173 | 169
  Pain: Post CYD vaccination 3: number analyzed (Participants) | 144 | 140
  Pain: Post CYD vaccination 3 | 65 | 59
  Erythema: Post any CYD/Cervarix vaccine: number analyzed (Participants) | 231 | 234
  Erythema: Post any CYD/Cervarix vaccine | 64 | 61
  Erythema: Post CYD/Cervarix vaccination 1: number analyzed (Participants) | 231 | 234
  Erythema: Post CYD/Cervarix vaccination 1 | 49 | 43
  Erythema: Post CYD/Cervarix vaccination 2: number analyzed (Participants) | 226 | 229
  Erythema: Post CYD/Cervarix vaccination 2 | 41 | 34
  Erythema: Post CYD vaccination 3: number analyzed (Participants) | 144 | 140
  Erythema: Post CYD vaccination 3 | 6 | 11
  Swelling: Post any CYD/Cervarix vaccine: number analyzed (Participants) | 231 | 234
  Swelling: Post any CYD/Cervarix vaccine | 73 | 60
  Swelling: Post CYD/Cervarix vaccination 1: number analyzed (Participants) | 231 | 234
  Swelling: Post CYD/Cervarix vaccination 1 | 55 | 44
  Swelling: Post CYD/Cervarix vaccination 2: number analyzed (Participants) | 226 | 229
  Swelling: Post CYD/Cervarix vaccination 2 | 48 | 35
  Swelling: Post CYD vaccination 3: number analyzed (Participants) | 144 | 139
  Swelling: Post CYD vaccination 3 | 8 | 10

11. Secondary Outcome: Number of Participants Reporting Solicited Systemic Reactions Following Vaccination With Cervarix or CYD Dengue Vaccine
Description: Solicited systemic reactions included Fever, Headache, Malaise, Myalgia, and Asthenia. At Visit 1 and Visit 4, participants from Group 1 received both Cervarix and CYD vaccination and participants from Group 2 received only Cervarix vaccination. At Visit 2 and Visit 5, only participants from Group 2 received CYD vaccination whereas the participants from Group 1 received no vaccination.
Time Frame: Up to 14 days after any and each vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 237 | 241
Participants
  Fever: Post any vaccination: number analyzed (Participants) | 230 | 234
  Fever: Post any vaccination | 25 | 35
  Fever: Post vaccination 1 (Visit 1): number analyzed (Participants) | 230 | 234
  Fever: Post vaccination 1 (Visit 1) | 14 | 8
  Fever: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 230
  Fever: Post CYD vaccination 1 (Visit 2) |  | 14
  Fever: Post vaccination 2 (Visit 4): number analyzed (Participants) | 216 | 228
  Fever: Post vaccination 2 (Visit 4) | 10 | 12
  Fever: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 227
  Fever: Post CYD vaccination 2 (Visit 5) |  | 8
  Fever: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 143 | 139
  Fever: Post CYD vaccination 3 (Visit 7) | 5 | 3
  Headache: Post any vaccination: number analyzed (Participants) | 231 | 234
  Headache: Post any vaccination | 101 | 111
  Headache: Post vaccination 1 (Visit 1): number analyzed (Participants) | 231 | 234
  Headache: Post vaccination 1 (Visit 1) | 83 | 69
  Headache: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 231
  Headache: Post CYD vaccination 1 (Visit 2) |  | 54
  Headache: Post vaccination 2 (Visit 4): number analyzed (Participants) | 226 | 229
  Headache: Post vaccination 2 (Visit 4) | 47 | 48
  Headache: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 227
  Headache: Post CYD vaccination 2 (Visit 5) |  | 36
  Headache: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 144 | 140
  Headache: Post CYD vaccination 3 (Visit 7) | 18 | 15
  Malaise: Post any vaccination: number analyzed (Participants) | 231 | 234
  Malaise: Post any vaccination | 113 | 133
  Malaise: Post vaccination 1 (Visit 1): number analyzed (Participants) | 231 | 234
  Malaise: Post vaccination 1 (Visit 1) | 84 | 84
  Malaise: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 231
  Malaise: Post CYD vaccination 1 (Visit 2) |  | 56
  Malaise: Post vaccination 2 (Visit 4): number analyzed (Participants) | 226 | 229
  Malaise: Post vaccination 2 (Visit 4) | 73 | 72
  Malaise: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 227
  Malaise: Post CYD vaccination 2 (Visit 5) |  | 47
  Malaise: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 144 | 140
  Malaise: Post CYD vaccination 3 (Visit 7) | 19 | 28
  Myalgia: Post any vaccination: number analyzed (Participants) | 231 | 234
  Myalgia: Post any vaccination | 160 | 168
  Myalgia: Post vaccination 1 (Visit 1): number analyzed (Participants) | 231 | 234
  Myalgia: Post vaccination 1 (Visit 1) | 129 | 124
  Myalgia: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 231
  Myalgia: Post CYD vaccination 1 (Visit 2) |  | 76
  Myalgia: Post vaccination 2 (Visit 4): number analyzed (Participants) | 226 | 229
  Myalgia: Post vaccination 2 (Visit 4) | 96 | 95
  Myalgia: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 227
  Myalgia: Post CYD vaccination 2 (Visit 5) |  | 60
  Myalgia: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 144 | 140
  Myalgia: Post CYD vaccination 3 (Visit 7) | 26 | 31
  Asthenia: Post any vaccination: number analyzed (Participants) | 231 | 234
  Asthenia: Post any vaccination | 93 | 95
  Asthenia: Post vaccination 1 (Visit 1): number analyzed (Participants) | 231 | 234
  Asthenia: Post vaccination 1 (Visit 1) | 72 | 53
  Asthenia: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 231
  Asthenia: Post CYD vaccination 1 (Visit 2) |  | 47
  Asthenia: Post vaccination 2 (Visit 4): number analyzed (Participants) | 226 | 229
  Asthenia: Post vaccination 2 (Visit 4) | 51 | 35
  Asthenia: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 227
  Asthenia: Post CYD vaccination 2 (Visit 5) |  | 30
  Asthenia: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 144 | 140
  Asthenia: Post CYD vaccination 3 (Visit 7) | 16 | 13

12. Secondary Outcome: Number of Participants Reporting Unsolicited AEs Following Vaccination With Cervarix or CYD Dengue Vaccine
Description: An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the CRF in terms of diagnosis and/or onset post-vaccination. At Visit 1 and Visit 4, participants from Group 1 received both Cervarix and CYD vaccination and participants from Group 2 received only Cervarix vaccination. At Visit 2 and Visit 5, only participants from Group 2 received CYD vaccination whereas the participants from Group 1 received no vaccination.
Time Frame: Up to 28 days after any and each vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 237 | 241
Participants
  Post any vaccination | 50 | 76
  Post vaccination 1 (Visit 1) | 33 | 37
  Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 233
  Post CYD vaccination 1 (Visit 2) |  | 25
  Post vaccination 2 (Visit 4): number analyzed (Participants) | 227 | 229
  Post vaccination 2 (Visit 4) | 26 | 23
  Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 228
  Post CYD vaccination 2 (Visit 5) |  | 15
  Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 145 | 141
  Post CYD vaccination 3 (Visit 7) | 5 | 5

13. Secondary Outcome: Number of Participants Reporting Non-serious Adverse Event of Special Interests (AESIs) Following Vaccination With Cervarix or CYD Dengue Vaccine
Description: AESI were AEs that were considered by the Sponsor to be relevant for the monitoring of the safety profile of the investigational vaccine.
Time Frame: Up to 7 days after any and each vaccination
Population: Analysis was performed on safety analysis set. Here, 'number analyzed' signifies participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 237 | 241
Participants
  Post any CYD/Cervarix vaccination | 0 | 0
  Post CYD/Cervarix vaccination 1 | 0 | 0
  Post CYD/Cervarix vaccination 2: number analyzed (Participants) | 227 | 229
  Post CYD/Cervarix vaccination 2 | 0 | 0
  Post CYD/Cervarix vaccination 3: number analyzed (Participants) | 145 | 141
  Post CYD/Cervarix vaccination 3 | 0 | 0

14. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Including Serious AESIs Following Vaccination With Cervarix or CYD Dengue Vaccine
Description: An SAEs were AEs resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or a medically important event. An AESIs were AEs that were considered by the Sponsor to be relevant for the monitoring of the safety profile of the investigational vaccine.
Time Frame: From Day 0 up to 6 months after the last CYD or Cervarix vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 237 | 241
Participants
  SAE | 6 | 0
  Serious AESI | 0 | 0

15. Secondary Outcome: Number of Participants Reporting Cases of Virologically Confirmed Dengue (VCD) Hospitalization Following Vaccination With Cervarix or CYD Dengue Vaccine
Description: Hospitalized suspected dengue case was defined as an acute febrile illness with diagnosis of dengue requiring hospitalization (with bed attribution). In such cases, 1 unplanned acute blood sample (within the first 5 days after fever onset) was collected for virological confirmation of hospitalized suspected dengue case. A suspected case was considered VCD if there was a detection of wild type dengue virus by dengue non-structural protein 1 antigen ELISA and/or dengue reverse transcriptase-polymerase chain reactions.
Time Frame: From Day 0 up to 6 months after the last CYD or Cervarix vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Cervarix (Concomitant Administration) | CYD Dengue Vaccine + Cervarix (Sequential Administration)
Number analyzed (Participants) | 237 | 241
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from Day 0 up to Day 28 post any vaccination. Solicited Reaction (SR) were collected from Day 0 up to Day 14 post vaccination. The SAEs were collected throughout the trial (up to Month 14), i.e,. 6 months after last CYD vaccination.
Description: The SR was an AE that was prelisted (i.e., solicited) in the electronic CRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was performed on safety analysis set.
Groups:
- CYD Dengue Vaccine + Cervarix (Sequential Administration): Participants received 3 doses of CYD dengue vaccine 0.5 mL SC at Day 0, Month 6, and Month 12 and 2 doses of Cervarix vaccine 0.5 mL IM concomitantly with the 2 first doses of CYD dengue vaccine.
- CYD Dengue Vaccine + Cervarix (Concomitant Administration): Participants received 3 doses of CYD dengue vaccine 0.5 mL SC at Month 1, Month 7, and Month 13 along with the 2 doses of Cervarix vaccine 0.5 mL IM at Day 0 and Month 6 sequentially (i.e., one month before) to each of the 2 first doses of CYD dengue vaccine.
Arm/Group | CYD Dengue Vaccine + Cervarix (Sequential Administration) | CYD Dengue Vaccine + Cervarix (Concomitant Administration)
All-Cause Mortality (participants affected / at risk) | 0/237 | 0/241
Serious Adverse Events (participants affected / at risk) | 6/237 | 0/241
Other Adverse Events (participants affected / at risk) | 222/237 | 228/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine + Cervarix (Sequential Administration) (N=237) | CYD Dengue Vaccine + Cervarix (Concomitant Administration) (N=241)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine + Cervarix (Sequential Administration) (N=237) | CYD Dengue Vaccine + Cervarix (Concomitant Administration) (N=241)
Asthenia (General disorders) | 93 (139) | 95 (178)
Injection Site Erythema (General disorders) | 64 (137) | 61 (116)
Injection Site Pain (General disorders) | 212 (659) | 221 (628)
Injection Site Swelling (General disorders) | 73 (154) | 60 (115)
Malaise (General disorders) | 113 (176) | 133 (287)
Pyrexia (General disorders) | 25 (29) | 37 (47)
Nasopharyngitis (Infections and infestations) | 8 (9) | 22 (26)
Pharyngitis (Infections and infestations) | 13 (13) | 20 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 160 (251) | 168 (386)
Headache (Nervous system disorders) | 102 (149) | 113 (227)

LIMITATIONS AND CAVEATS:
Change of population for non-inferiority reduced to dengue seropositive participants and time window for vaccination not reached (study hold), hence non-inferiority analysis not performed & immunogenicity analysis was performed on FAS & not on PPS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02979535/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT02979535/SAP_000.pdf